CLINICAL TRIAL: NCT05100472
Title: Phase II Trial of Short Course Androgen Deprivation, Hypofractionated Pelvic Radiation and a Brachytherapy Boost for NCCN High-Risk Prostate Cancer With Low-Intermediate Risk Decipher Genomic Score
Brief Title: A Study of Shorter Course Hormone Therapy and Radiation for High-risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-405
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Hypofractionated Pelvic Radiation; Brachytherapy Boost; NCCN High-Risk Prostate Cancer; Low-Intermediate Risk Decipher Genomic Score; Androgen Deprivation; 21-405
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Brachytherapy

STUDY DESIGN:
Intervention Model Description: This is a phase II single arm trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hormone Therapy and Radiation (Experimental): Patients enrolled in this study will receive ADT for 6 months which will consist of bicalutamide 50 mg PO daily starting approximately 1-2 weeks before leuprolide 22.5mg injected every 3 months. The HDR prostate brachytherapy procedure will be performed approximately 3 months after starting ADT to allow for potential radiosensitization and cytoreduction. Approximately 4 weeks after the HDR boost, patients will receive image-guided, intensity-modulated, hypofractionated radiation therapy targeting the prostate, seminal vesicles and pelvic lymph nodes to a dose of 25 Gy in 5 fractions delivered daily.
  Interventions: Biological: Androgen deprivation therapy (ADT); Radiation: Brachytherapy; Radiation: Hypofractionated pelvic External beam radiation

INTERVENTIONS:
Biological: Androgen deprivation therapy (ADT) — ADT will include bicalutamide 50 mg PO daily started 1-2 weeks before leuprolide 22.5mg IM or SQ delivered every 3 months x 2. Bicalutamide will be continued through radiation and then discontinued on the day of the last fraction. Leuprolide can be given at different doses, but must be given for a total planned duration of 6 months.
Radiation: Brachytherapy — After approximately 3 months (+/- 1 month) of neoadjuvant ADT, patients will undergo general anesthesia for outpatient transperineal high dose rate (HDR) interstitial prostate brachytherapy implant.
Radiation: Hypofractionated pelvic External beam radiation — Patients will receive image-guided, intensity-modulated, hypofractionated radiation therapy targeting the prostate, seminal vesicles and pelvic lymph nodes to a dose of 25 Gy in 5 fractions delivered daily.

SUMMARY:
The purpose of this study is to find out whether combining a shorter than standard course of ADT with standard prostate brachytherapy and hypofractionated external beam radiation therapy is a safe and effective way to prevent high-risk prostate cancer from coming back and/or spreading to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-proven diagnosis of prostate adenocarcinoma
* Clinical stage T3-4 or Gleason score 8-10 or PSA >20 ng/ml

  °If radiographic T3-T4 is the only high-risk factor, it must be "consistent with" or >90% probability of having T3-T4 disease determined by the reading radiologist.
* Decipher genomic score ≤0.6
* Willing and able to provide written informed consent and Authorization for Use and Release of Health and Research Study Information (HIPAA authorization)
* Age ≥18
* KPS ≥70 or ECOG 0-2
* Estimated life expectancy >5 years
* Baseline prostate volume ≤90 cc
* Baseline IPSS ≤20
* No contraindications to ADT, brachytherapy, or pelvic external beam radiation therapy as determined by the treating radiation oncologist per standard practice
* Patients who have already started ADT consisting of bicalutamide 50 mg PO daily with leuprolide or an equivalent GnRH analogue are eligible if given for ≤ 60 days prior to registration

Exclusion Criteria:

* Regional lymph node or metastatic disease
* Prior pelvic radiation
* Prior prostate surgery (including TURP or cryosurgery)
* Prior history of inflammatory bowel disease
* Unable to undergo anesthesia or brachytherapy
* Active second malignancy or past history of malignancies diagnosed within the last 2 years that requires active therapy and/or in remission, with the exception of resected non-melanoma skin cancers, non-muscle invasive bladder cancer, stage I head and neck cancer, or stage I colorectal cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 50 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Distant metastatic disease-free (DMF) rate | 3 years
  Time to distant metastases will be estimated from the date of enrollment until distant metastases

SECONDARY OUTCOMES:
Pathological response rate | Between 24-36 months after radiation
Cumulative incidence of biochemical failure | 3 years
Overall survival rate | 3 years
Acute and late physician-scored toxicity | 3 years
  Using CTCAE v5.0. NCI Common Toxicity Criteria. The NCI scales are simple to complete and provide a means for assessing patient symptoms. Only the CTCAE v 5.0 will be used in toxicity grading.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gorovets, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm